CLINICAL TRIAL: NCT05936697
Title: Neurofeedback Training to Improve Prefrontal Functioning in Older Adults With Subclinical Depression and Anxiety: a Randomised Control Trial
Brief Title: Neurofeedback Training For Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20221103002
Record Dates: First submitted 2023-04-16; First posted 2023-07-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: Depression, Anxiety
Keywords: Neurofeedback; Prefrontal Cortex
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: The participants will be randomly and equally assigned to one of three neurofeedback training groups: (1) sham, (2) EEG, and (3) fNIRS. Each participant will complete a neurophysiological assessment (1) before, (2) immediately after, and (3) 1 month after the intervention.
Who Masked: Participant, Investigator
Masking Description: During each training session, a cap adjusted to the participant's head size will be used to mount the EEG and fNIRS sensors. The hardware setup will be the same for all groups to ensure that both the participant and the experimenter are blinded to the training group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Group (Sham Comparator): During training, participants will be asked to follow the instructions on a computer screen and complete five rounds of task. Each round starts with a 30-s rest phase followed by 4.5 min of self-regulation phase. At the rest phase, a fixed cross will appear onscreen, and participants will be instructed to sit still and relax. At the regulation phase, they will be asked to make the person smile (as an intrinsic social reward) but without tips. The intensity of smiling will be manipulated by morphing photographs of a neutral and a happy face and will represent the increase in either frontal alpha asymmetry or frontal oxyhaemoglobin asymmetry. The values at the moment will be compared against the baseline. Participants will undergo a 3-min rest period before and after each training session to track changes in resting-state brain activity. In the sham condition, participants will receive visual feedback based on pre-recordings and/or other participants' recordings.
  Interventions: Other: Baseline Training
- fNIRS Group (Experimental): During training, participants will be asked to follow the instructions on a computer screen and complete five rounds of task. Each round starts with a 30-s rest phase followed by 4.5 min of self-regulation phase. At the rest phase, a fixed cross will appear onscreen, and participants will be instructed to sit still and relax. At the regulation phase, they will be asked to make the person smile (as an intrinsic social reward) but without tips. The intensity of smiling will be manipulated by morphing photographs of a neutral and a happy face and will represent the increase in either frontal alpha asymmetry or frontal oxyhaemoglobin asymmetry. The values at the moment will be compared against the baseline. Participants will undergo a 3-min rest period before and after each training session to track changes in resting-state brain activity. In the fNIRS condition, participants will receive visual feedback based on their own fNIRS recordings.
  Interventions: Device: fNIRS
- EEG Group (Experimental): During training, participants will be asked to follow the instructions on a computer screen and complete five rounds of task. Each round starts with a 30-s rest phase followed by 4.5 min of self-regulation phase. At the rest phase, a fixed cross will appear onscreen, and participants will be instructed to sit still and relax. At the regulation phase, they will be asked to make the person smile (as an intrinsic social reward) but without tips. The intensity of smiling will be manipulated by morphing photographs of a neutral and a happy face and will represent the increase in either frontal alpha asymmetry or frontal oxyhaemoglobin asymmetry. The values at the moment will be compared against the baseline. Participants will undergo a 3-min rest period before and after each training session to track changes in resting-state brain activity. In the EEG condition, participants will receive visual feedback based on their own EEG recordings.
  Interventions: Device: EEG

INTERVENTIONS:
Device: fNIRS — For fNIRS to be recorded by the wearable OctaMon+ system (Artinis Medical Systems, The Netherlands), two sources, each surrounded by four detectors positioned approximately 3 cm apart, will be placed on the scalp such that the two channels near the fissure on each side of the head are surrounded F3 and F4. Data will be sampled at 50 Hz.
  Arms: fNIRS Group
Device: EEG — For EEG to be recorded by the ANT eego rt8 amplifier (ANT Neuro, Hengelo, The Netherlands), electrodes will be placed at Fp1, F3, F4, Fz, Fpz, Cz, GND (ground), lower VEOG, and on the two earlobes (references). Data will be collected at 2,048 Hz.
  Arms: EEG Group
Other: Baseline Training — In the sham condition, participants will receive visual feedback based on pre-recordings and/or other participants' recordings. Participants will undergo a 3-min rest period before and after each training session to track changes in resting-state brain activity within and across sessions.
  Arms: Sham Group

SUMMARY:
Symptoms of depression and anxiety are common in older adults and are associated with poor outcomes and the risk of dementia. The prefrontal cortex (PFC) is crucial for emotion regulation. Poor PFC function may underlie subclinical depression and anxiety symptoms in older people, which could progress to clinical conditions. Neurofeedback training based on electroencephalography (EEG) or functional near-infrared spectroscopy (fNIRS) teaches individuals to self-regulate different aspects of brain activity and induce neurocognitive improvements. This proposed project will examine whether prefrontal EEG and fNIRS neurofeedback training programmes can enhance the mood and cognition of older adults with subclinical depression and anxiety.

DETAILED DESCRIPTION:
Background:

Subclinical symptoms of depression and anxiety are common in older adults, with some estimates indicating that these symptoms are present in 10-52% of community-dwelling older adults. Some studies have shown that older adults with subclinical depression and anxiety are more likely than those with low levels of relevant symptoms to be diagnosed with affective disorders and mild cognitive impairment or dementia later in life. Thus, interventions for older people with elevated subclinical symptoms of depression and anxiety are crucial for preventing affective disorders and dementia late in life. During negative emotional experiences, the prefrontal cortex (PFC) plays a pivotal role in downregulating activity. PFC dysfunction may cause different mood and anxiety symptoms.

Neurofeedback training is a non-pharmaceutical neurorehabilitation technique that can potentially improve prefrontal function and enhance mental health and cognitive functions. This technique uses sensory feedback to teach individuals to self-regulate specific brain activities, with the goal of inducing long-term neuroplasticity and functional improvements. Traditionally, neurofeedback training has been conducted using EEG, and much research has applied such training interventions for the treatment of a variety of psychiatric disorders. In recent years, interest in using fNIRS to deliver neurofeedback training has grown. The underlying mechanism of such training with fNIRS is different from that of training with EEG. Compared with EEG, fNIRS has a lower temporal resolution but a higher spatial resolution and is more resilient to movement artifacts. In addition, one recent study showed that patients with social anxiety disorder had reduced anxiety symptoms after fNIRS neurofeedback training.

Research Plan and Methodology:

Design: This proposed project has been designed in accordance with current consensus on the reporting and experimental design of clinical and cognitive-behavioural neurofeedback studies. The participants will be randomly and equally assigned to one of three neurofeedback training groups: (1) sham, (2) EEG, and (3) fNIRS. Each participant will complete a neurophysiological assessment (1) before, (2) immediately after, and (3) 1 month after intervention.

Participants: 90 older adults without dementia will be recruited via advertisements at PolyU and NGOs. The inclusion criteria is: (i) age of 60-79 years; (ii) right-handedness as assessed using the short form of the Edinburgh Handedness Inventory; (iii) a moderate or higher score on at least one of the depression and anxiety subscales (but not necessarily both) of the Depression Anxiety Stress Scale-21 (DASS-21); (iv) no history of neurological or psychiatric disorder; (iv) no history of traumatic brain injury requiring hospitalisation; (vi) not currently using psychotropic medication; (vii) ability to read Traditional Chinese; (viii) normal or corrected-to-normal vision; and (ix) a score of at least 19 on the Hong Kong Montreal Cognitive Assessment (HK-MoCA).

The inclusion criteria that the investigators planned to use were based on those employed by prefrontal neurofeedback studies in mood or anxiety disorders. Conventionally, participants are selected based on a certain threshold of depressive or anxiety symptoms, neither cognitive nor brain dysfunction constitutes an inclusion criterion. Nevertheless, since variation in cognitive and PFC functioning levels may affect the treatment response, subsequent analyses will consider baseline cognitive and PFC functioning levels.

Study Procedures: Potential participants will first be subjected to a screening evaluation to assess eligibility. Eligible individuals will be invited to PolyU for assessment and training. The training will comprise 10 60-min sessions conducted within 4 weeks. Each session will include 25-min effective training time, for a total training time of 250 min, in keeping with recent recommendations. In addition, the participants will undertake 3 experimental tasks under simultaneous EEG-fNIRS recording and complete several questionnaires at 3 time points, as described in the 'Neurophysiological Assessment' section. Multiple studies have demonstrated that EEG, fNIRS, and neurofeedback training can be applied to older adults over 70, and even to individuals with dementia. Therefore, the investigators expect that older adults who are screened for dementia by the HK-MoCA will be able to follow both the assessment and training protocols.

Neurofeedback Training: During training, participants will be asked to follow the instructions on a computer screen. They will complete five rounds of training task. Each round starts with a 30-s rest phase followed by 4.5 min of self-regulation phase. During the rest phase, a fixation cross will appear onscreen, and the participants will be instructed to sit still and relax. During the regulation period, the participants will be asked to make the square change from white to black (i.e., an intrinsic social reward) but will not be given specific strategies. The darkness of colour will represent the increase in either frontal alpha asymmetry or frontal oxyhaemoglobin (HbO) asymmetry. The values at the moment will be compared against the 20-s pre-regulation baseline. In the sham condition, participants will receive visual feedback based on pre-recordings and/or other participants' recordings. Participants will undergo a 3-min rest period before and after each training session to track changes in resting-state brain activity within and across sessions.

During each training session, a cap adjusted to the participant's head size will be used to mount the EEG and fNIRS sensors. The hardware setup will be the same for all groups to ensure that both the participant and the experimenter are blinded. For EEG to be recorded by the ANT eego rt8 amplifier (ANT Neuro, Hengelo, The Netherlands), electrodes will be placed at Fp1, F3, F4, Fz, Fpz, Cz, GND (ground), lower VEOG, and on the two earlobes (references). Data will be collected at 2,048 Hz. For fNIRS to be recorded by the wearable OctaMon+ system (Artinis Medical Systems, Gelderland, The Netherlands), two sources, each surrounded by four detectors positioned approximately 3 cm apart, will be placed on the scalp such that the two channels near the cerebral fissure on each side of the hemispheres are surrounded F3 and F4. Data will be sampled at 50 Hz. Depending on the training group, frontal asymmetry in terms of the difference in alpha power (8-13 Hz) between F3 and F4 and the mean change in HbO concentration between the left and right PFC will be chosen as the target objective. For both real training groups, real-time data streaming will be performed using the Lab Streaming Layer and OpenVibe according to published guidelines.

Neurophysiological Assessment: A 1.5-h neurophysiological assessment will be administered at each of 3 time points (pre, post, and 1-month follow-up) to evaluate the effects of neurofeedback training. The participants will complete the DASS-21 (Chinese version) to measure their depressive and anxiety symptoms over the last week; the Hospital Anxiety and Depression Scale (HADS; Chinese version) to measure their signs of anxiousness and depression during the previous week; the Pittsburgh Sleep Quality Index to measure their sleep quality over the last month; the Satisfaction with Life Scale (Chinese version) to quantify their general life satisfaction; and Lawton Instrumental Activities of Daily Living Scale (IADL; Chinese version) to assess independent living skills. The participants will also complete three computerised tasks to assess different components of frontal cognitive function under simultaneous EEG-fNIRS measurements, using the same setup as neurofeedback training. At the first visit, the participants will also complete the HK-MoCA to screen for dementia. Immediately after the intervention, they will be asked whether they know their treatment group assignment to check the strength of blinding.

Each assessment task (eyes open, Emotional Stroop, n-back) proposed for this research will comprise a difficult and an easy condition. The eyes open test is used to let the machine measure the activation baseline when the participants open their eyes. It requires participants to maintain their eyes open for 3 minutes. The Emotional Stroop task is used to assess inhibitory control. Participants are shown photos of different emotions with unrelated traditional Chinese emotion names. They are asked to name the photos by emotion. It requires participants to inhibit their emotions lead by the wordings and react to the content of the photo. Differences in accuracy and mean reaction time (RT) and changes in the prefrontal HbO concentration and theta power between the two conditions will be the dependent variables. The n-back task is used to assess working memory. During the task, participants are shown a sequence of digits and asked to judge via button press whether the digit they are seeing is zero (0-back; easy) or the same as the digit they saw two trials before (2-back; difficult). Differences in accuracy and mean RT and changes in the prefrontal HbO concentration and theta power between the two conditions will be the dependent variables.

Data Analysis: In this project, the primary outcome measures are mood and anxiety measures (i.e., DASS-21 and HADS scores), and the secondary outcome measures are task performance and PFC measures, as well as other mental health measures. The outcome measures will be analysed according to the CRED-nf checklist. Linear mixed models with group (sham, EEG, fNIRS), time (baseline, post, follow-up), and condition (easy, difficult) as the fixed factors; and the subject as a random factor will be used to analyse the behavioural, fNIRS, and EEG data. The investigators expect that participants in the two real neurofeedback training groups will demonstrate significant improvements in mental health, cognitive function, and frontal lobe function at the post and follow-up assessments relative to the sham group participants. In addition, the investigators will evaluate differences in pre-post changes in mental health and cognitive functions between the two real training groups. Moreover, the investigators will examine the correlation between baseline cognitive and PFC functioning levels and the pre-post changes in DASS-21 scores to elucidate individual differences in the treatment response for each neurofeedback group.

ELIGIBILITY:
Inclusion Criteria:

* (i) age of 60-79 years;
* (ii) right-handedness as assessed using the short form of the Edinburgh Handedness Inventory (Veale, 2014);
* (iii) a moderate or higher score on at least one of the depression and anxiety subscales (but not necessarily both) of the Depression Anxiety Stress Scale-21 (DASS-21), which has been shown to yield reliable and valid scores;
* (iv) no history of neurological or psychiatric disorder;
* (v) no history of traumatic brain injury requiring hospitalisation;
* (vi) not currently using psychotropic medication;
* (vii) ability to read Traditional Chinese text;
* (viii) normal or corrected-to-normal vision; and
* (ix) a score of at least 19 on the Hong Kong Montreal Cognitive Assessment

Exclusion Criteria:

* does not fulfill any of the above criteria

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Mood symptoms (post) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in the HADS depression score (The Hospital Anxiety and Depression Scale (HADS) depression score has a minimum value of 0 and a maximum value of 21. Higher scores indicate a worse outcome. A score of 0-7 indicates normal, 8-10 indicates mild depression, 11-14 indicates borderline depression, and 15-21 indicates depression.)
Mood symptoms (follow-up) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in the HADS depression score at follow up (The Hospital Anxiety and Depression Scale (HADS) depression score has a minimum value of 0 and a maximum value of 21. Higher scores indicate a worse outcome. A score of 0-7 indicates normal, 8-10 indicates mild depression, 11-14 indicates borderline depression, and 15-21 indicates depression.)
Anxiety symptoms (post) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in the HADS anxiety score (The Hospital Anxiety and Depression Scale (HADS) anxiety score has a minimum value of 0 and a maximum value of 21. Higher scores indicate a worse outcome. A score of 0-7 indicates normal, 8-10 indicates mild anxiety, 11-14 indicates borderline anxiety, and 15-21 indicates anxiety.)
Anxiety symptoms (follow-up) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in the HADS anxiety score at follow-up (The Hospital Anxiety and Depression Scale (HADS) anxiety score has a minimum value of 0 and a maximum value of 21. Higher scores indicate a worse outcome. A score of 0-7 indicates normal, 8-10 indicates mild anxiety, 11-14 indicates borderline anxiety, and 15-21 indicates anxiety.)

SECONDARY OUTCOMES:
Stroop (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Stroop mean reaction time
Stroop (follow-up; RT) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in Stroop mean reaction time at follow-up
Stroop (post; accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in Stroop accuracy
Stroop (follow-up; accuracy) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in Stroop accuracy at follow-up
Stroop (post; fNIRS) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in mean change in oxyhemoglobin concentration measured by fNIRS
Stroop (follow-up; fNIRS) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in mean change in oxyhemoglobin concentration measured by fNIRS at follow-up
Stroop (post; EEG) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in stimulus-locked N450 amplitude measured by EEG
Stroop (follow-up; EEG) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in stimulus-locked N450 amplitude measured by EEG at follow-up
n-back (post; RT) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in n-back mean reaction time
n-back (follow-up; RT) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in n-back mean reaction time at follow-up
n-back (post; accuracy) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in n-back accuracy
n-back (follow-up; accuracy) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in n-back accuracy at follow-up
n-back (post; fNIRS) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in mean change in oxyhemoglobin concentration measured by fNIRS
n-back (follow-up; fNIRS) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in mean change in oxyhemoglobin concentration measured by fNIRS at follow-up
n-back (post; EEG) | Within 1 week before the first training session, and within 1 week after the last training session
  Change in stimulus-locked P300 amplitude measured by EEG at follow-up
n-back (follow-up; EEG) | Within 1 week before the first training session, and within 1 month after the last training session
  Change in stimulus-locked P300 amplitude measured by EEG at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kin Chung Michael Yeung, Study Chair — The Education University of Hong Kong
Locations (1):
- Faculty of Health and Social Sciences OF The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Personal information obtained for this study will be kept totally secret, and each participant will be assigned a unique serial number. We will properly secure their identity and privacy, as well as the personal data of all participants. The Confidentiality and Privacy Ordinance of The Hong Kong Polytechnic University shall protect and keep all medical data. Personal information will be stored in an encrypted file with just a code number to identify it. All personal data will be removed five years after the study project is completed. Research findings may be published in international academic publications or at conferences, but all personal information will be kept confidential.

REFERENCES:
- [Background] Flint AJ, Rifat SL. Factor structure of the hospital anxiety and depression scale in older patients with major depression. Int J Geriatr Psychiatry. 2002 Feb;17(2):117-23. doi: 10.1002/gps.535. PMID 11813272
- [Background] Gomez, R., Summers, M., Summers, A., Wolf, A., & Summers, J. J. (2014). Depression Anxiety Stress Scales-21: Factor structure and test-retest invariance, and temporal stability and uniqueness of latent factors in older adults. Journal of Psychopathology and Behavioral Assessment, 36(2), 308-317.
- [Background] Norton PJ. Depression Anxiety and Stress Scales (DASS-21): psychometric analysis across four racial groups. Anxiety Stress Coping. 2007 Sep;20(3):253-65. doi: 10.1080/10615800701309279. PMID 17999228
- [Background] Veale JF. Edinburgh Handedness Inventory - Short Form: a revised version based on confirmatory factor analysis. Laterality. 2014;19(2):164-77. doi: 10.1080/1357650X.2013.783045. Epub 2013 May 10. PMID 23659650
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Adolph D, Margraf J. The differential relationship between trait anxiety, depression, and resting frontal alpha-asymmetry. J Neural Transm (Vienna). 2017 Mar;124(3):379-386. doi: 10.1007/s00702-016-1664-9. Epub 2016 Dec 16. PMID 27987054
- [Background] Barry RJ, De Blasio FM. EEG differences between eyes-closed and eyes-open resting remain in healthy ageing. Biol Psychol. 2017 Oct;129:293-304. doi: 10.1016/j.biopsycho.2017.09.010. Epub 2017 Sep 21. PMID 28943465
- [Background] Beaudreau SA, O'Hara R. Late-life anxiety and cognitive impairment: a review. Am J Geriatr Psychiatry. 2008 Oct;16(10):790-803. doi: 10.1097/JGP.0b013e31817945c3. PMID 18827225
- [Background] Beekman AT, de Beurs E, van Balkom AJ, Deeg DJ, van Dyck R, van Tilburg W. Anxiety and depression in later life: Co-occurrence and communality of risk factors. Am J Psychiatry. 2000 Jan;157(1):89-95. doi: 10.1176/ajp.157.1.89. PMID 10618018
- [Background] Bruder GE, Stewart JW, McGrath PJ. Right brain, left brain in depressive disorders: Clinical and theoretical implications of behavioral, electrophysiological and neuroimaging findings. Neurosci Biobehav Rev. 2017 Jul;78:178-191. doi: 10.1016/j.neubiorev.2017.04.021. Epub 2017 Apr 23. PMID 28445740
- [Background] Bryant C, Jackson H, Ames D. The prevalence of anxiety in older adults: methodological issues and a review of the literature. J Affect Disord. 2008 Aug;109(3):233-50. doi: 10.1016/j.jad.2007.11.008. Epub 2007 Dec 26. PMID 18155775
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cui X, Bray S, Reiss AL. Functional near infrared spectroscopy (NIRS) signal improvement based on negative correlation between oxygenated and deoxygenated hemoglobin dynamics. Neuroimage. 2010 Feb 15;49(4):3039-46. doi: 10.1016/j.neuroimage.2009.11.050. Epub 2009 Nov 26. PMID 19945536
- [Background] Cuijpers P, Koole SL, van Dijke A, Roca M, Li J, Reynolds CF 3rd. Psychotherapy for subclinical depression: meta-analysis. Br J Psychiatry. 2014 Oct;205(4):268-74. doi: 10.1192/bjp.bp.113.138784. PMID 25274315
- [Background] Delpy DT, Cope M, van der Zee P, Arridge S, Wray S, Wyatt J. Estimation of optical pathlength through tissue from direct time of flight measurement. Phys Med Biol. 1988 Dec;33(12):1433-42. doi: 10.1088/0031-9155/33/12/008. PMID 3237772
- [Background] Ehlis, A. C., Barth, B., Hudak, J., Storchak, H., Weber, L., Kimmig, A. C. S., ... & Fallgatter, A. J. (2018). Near-infrared spectroscopy as a new tool for neurofeedback training: Applications in psychiatry and methodological considerations. Japanese Psychological Research, 60(4), 225-241.
- [Background] Etkin A, Buchel C, Gross JJ. The neural bases of emotion regulation. Nat Rev Neurosci. 2015 Nov;16(11):693-700. doi: 10.1038/nrn4044. PMID 26481098
- [Background] Fernandez-Alvarez J, Grassi M, Colombo D, Botella C, Cipresso P, Perna G, Riva G. Efficacy of bio- and neurofeedback for depression: a meta-analysis. Psychol Med. 2022 Jan;52(2):201-216. doi: 10.1017/S0033291721004396. Epub 2021 Nov 15. PMID 34776024
- [Background] Grahek I, Shenhav A, Musslick S, Krebs RM, Koster EHW. Motivation and cognitive control in depression. Neurosci Biobehav Rev. 2019 Jul;102:371-381. doi: 10.1016/j.neubiorev.2019.04.011. Epub 2019 May 27. PMID 31047891
- [Background] Haigh EAP, Bogucki OE, Sigmon ST, Blazer DG. Depression Among Older Adults: A 20-Year Update on Five Common Myths and Misconceptions. Am J Geriatr Psychiatry. 2018 Jan;26(1):107-122. doi: 10.1016/j.jagp.2017.06.011. Epub 2017 Jun 16. PMID 28735658
- [Background] Hammond, D. C. (2005). Neurofeedback treatment of depression and anxiety. Journal of Adult Development, 12(2), 131-137.
- [Background] Hammond, D. C. (2011). What is neurofeedback: An update. Journal of Neurotherapy, 15(4), 305-336.
- [Background] Imbir KK, Duda-Golawska J, Pastwa M, Sobieszek A, Wielgopolan A, Jankowska M, Modzelewska A, Zygierewicz J. Inhibitory control effectiveness can be improved: The role of arousal, subjective significance and origin of words in modified Emotional Stroop Test. PLoS One. 2022 Jun 28;17(6):e0270558. doi: 10.1371/journal.pone.0270558. eCollection 2022. PMID 35763510
- [Background] Kimmig AS, Dresler T, Hudak J, Haeussinger FB, Wildgruber D, Fallgatter AJ, Ehlis AC, Kreifelts B. Feasibility of NIRS-based neurofeedback training in social anxiety disorder: behavioral and neural correlates. J Neural Transm (Vienna). 2019 Sep;126(9):1175-1185. doi: 10.1007/s00702-018-1954-5. Epub 2018 Nov 29. PMID 30498952
- [Background] Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb;5(2):e45. doi: 10.1371/journal.pmed.0050045. PMID 18303940
- [Background] Kober SE, Spork R, Bauernfeind G, Wood G. Age-related differences in the within-session trainability of hemodynamic parameters: a near-infrared spectroscopy-based neurofeedback study. Neurobiol Aging. 2019 Sep;81:127-137. doi: 10.1016/j.neurobiolaging.2019.05.022. Epub 2019 Jun 5. PMID 31280116
- [Background] Kohl SH, Mehler DMA, Luhrs M, Thibault RT, Konrad K, Sorger B. The Potential of Functional Near-Infrared Spectroscopy-Based Neurofeedback-A Systematic Review and Recommendations for Best Practice. Front Neurosci. 2020 Jul 21;14:594. doi: 10.3389/fnins.2020.00594. eCollection 2020. PMID 32848528
- [Background] Kothe, C. (2014a). Lab Streaming Layer (LSL). Available online at: https://code.google.com/p/labstreaminglayer/
- [Background] Laborda-Sanchez F, Cansino S. The Effects of Neurofeedback on Aging-Associated Cognitive Decline: A Systematic Review. Appl Psychophysiol Biofeedback. 2021 Mar;46(1):1-10. doi: 10.1007/s10484-020-09497-6. Epub 2021 Jan 2. PMID 33389281
- [Background] Laborde-Lahoz P, El-Gabalawy R, Kinley J, Kirwin PD, Sareen J, Pietrzak RH. Subsyndromal depression among older adults in the USA: prevalence, comorbidity, and risk for new-onset psychiatric disorders in late life. Int J Geriatr Psychiatry. 2015 Jul;30(7):677-85. doi: 10.1002/gps.4204. Epub 2014 Oct 23. PMID 25345806
- [Background] Lee YJ, Kim HG, Cheon EJ, Kim K, Choi JH, Kim JY, Kim JM, Koo BH. The Analysis of Electroencephalography Changes Before and After a Single Neurofeedback Alpha/Theta Training Session in University Students. Appl Psychophysiol Biofeedback. 2019 Sep;44(3):173-184. doi: 10.1007/s10484-019-09432-4. PMID 30903394
- [Background] Li K, Jiang Y, Gong Y, Zhao W, Zhao Z, Liu X, Kendrick KM, Zhu C, Becker B. Functional near-infrared spectroscopy-informed neurofeedback: regional-specific modulation of lateral orbitofrontal activation and cognitive flexibility. Neurophotonics. 2019 Apr;6(2):025011. doi: 10.1117/1.NPh.6.2.025011. Epub 2019 Jun 8. PMID 31930153
- [Background] Marzbani H, Marateb HR, Mansourian M. Neurofeedback: A Comprehensive Review on System Design, Methodology and Clinical Applications. Basic Clin Neurosci. 2016 Apr;7(2):143-58. doi: 10.15412/J.BCN.03070208. PMID 27303609
- [Background] Mathersul D, Williams LM, Hopkinson PJ, Kemp AH. Investigating models of affect: relationships among EEG alpha asymmetry, depression, and anxiety. Emotion. 2008 Aug;8(4):560-72. doi: 10.1037/a0012811. PMID 18729586
- [Background] Meeks TW, Vahia IV, Lavretsky H, Kulkarni G, Jeste DV. A tune in "a minor" can "b major": a review of epidemiology, illness course, and public health implications of subthreshold depression in older adults. J Affect Disord. 2011 Mar;129(1-3):126-42. doi: 10.1016/j.jad.2010.09.015. PMID 20926139
- [Background] Mochcovitch MD, da Rocha Freire RC, Garcia RF, Nardi AE. A systematic review of fMRI studies in generalized anxiety disorder: evaluating its neural and cognitive basis. J Affect Disord. 2014;167:336-42. doi: 10.1016/j.jad.2014.06.041. Epub 2014 Jul 2. PMID 25020268
- [Background] Peeters F, Oehlen M, Ronner J, van Os J, Lousberg R. Neurofeedback as a treatment for major depressive disorder--a pilot study. PLoS One. 2014 Mar 18;9(3):e91837. doi: 10.1371/journal.pone.0091837. eCollection 2014. PMID 24642756
- [Background] Richard E, Reitz C, Honig LH, Schupf N, Tang MX, Manly JJ, Mayeux R, Devanand D, Luchsinger JA. Late-life depression, mild cognitive impairment, and dementia. JAMA Neurol. 2013 Mar 1;70(3):374-82. doi: 10.1001/jamaneurol.2013.603. PMID 23599941
- [Background] Renard, Y., Lotte, F., Gibert, G., Congedo, M., Maby, E., Delannoy, V., ... & Lécuyer, A. (2010). Openvibe: An open-source software platform to design, test, and use brain-computer interfaces in real and virtual environments. Presence, 19(1), 35-53.
- [Background] Ros T, Enriquez-Geppert S, Zotev V, Young KD, Wood G, Whitfield-Gabrieli S, Wan F, Vuilleumier P, Vialatte F, Van De Ville D, Todder D, Surmeli T, Sulzer JS, Strehl U, Sterman MB, Steiner NJ, Sorger B, Soekadar SR, Sitaram R, Sherlin LH, Schonenberg M, Scharnowski F, Schabus M, Rubia K, Rosa A, Reiner M, Pineda JA, Paret C, Ossadtchi A, Nicholson AA, Nan W, Minguez J, Micoulaud-Franchi JA, Mehler DMA, Luhrs M, Lubar J, Lotte F, Linden DEJ, Lewis-Peacock JA, Lebedev MA, Lanius RA, Kubler A, Kranczioch C, Koush Y, Konicar L, Kohl SH, Kober SE, Klados MA, Jeunet C, Janssen TWP, Huster RJ, Hoedlmoser K, Hirshberg LM, Heunis S, Hendler T, Hampson M, Guggisberg AG, Guggenberger R, Gruzelier JH, Gobel RW, Gninenko N, Gharabaghi A, Frewen P, Fovet T, Fernandez T, Escolano C, Ehlis AC, Drechsler R, Christopher deCharms R, Debener S, De Ridder D, Davelaar EJ, Congedo M, Cavazza M, Breteler MHM, Brandeis D, Bodurka J, Birbaumer N, Bazanova OM, Barth B, Bamidis PD, Auer T, Arns M, Thibault RT. Consensus on the reporting and experimental design of clinical and cognitive-behavioural neurofeedback studies (CRED-nf checklist). Brain. 2020 Jun 1;143(6):1674-1685. doi: 10.1093/brain/awaa009. PMID 32176800
- [Background] Shibasaki H. Human brain mapping: hemodynamic response and electrophysiology. Clin Neurophysiol. 2008 Apr;119(4):731-43. doi: 10.1016/j.clinph.2007.10.026. Epub 2008 Jan 9. PMID 18187361
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Snyder HR. Major depressive disorder is associated with broad impairments on neuropsychological measures of executive function: a meta-analysis and review. Psychol Bull. 2013 Jan;139(1):81-132. doi: 10.1037/a0028727. Epub 2012 May 28. PMID 22642228
- [Background] Snyder HR, Miyake A, Hankin BL. Advancing understanding of executive function impairments and psychopathology: bridging the gap between clinical and cognitive approaches. Front Psychol. 2015 Mar 26;6:328. doi: 10.3389/fpsyg.2015.00328. eCollection 2015. PMID 25859234
- [Background] Steenland K, Karnes C, Seals R, Carnevale C, Hermida A, Levey A. Late-life depression as a risk factor for mild cognitive impairment or Alzheimer's disease in 30 US Alzheimer's disease centers. J Alzheimers Dis. 2012;31(2):265-75. doi: 10.3233/JAD-2012-111922. PMID 22543846
- [Background] Steingrimsson S, Bilonic G, Ekelund AC, Larson T, Stadig I, Svensson M, Vukovic IS, Wartenberg C, Wrede O, Bernhardsson S. Electroencephalography-based neurofeedback as treatment for post-traumatic stress disorder: A systematic review and meta-analysis. Eur Psychiatry. 2020 Jan 31;63(1):e7. doi: 10.1192/j.eurpsy.2019.7. PMID 32093790
- [Background] Szymkowicz SM, Woods AJ, Dotson VM, Porges EC, Nissim NR, O'Shea A, Cohen RA, Ebner NC. Associations between subclinical depressive symptoms and reduced brain volume in middle-aged to older adults. Aging Ment Health. 2019 Jul;23(7):819-830. doi: 10.1080/13607863.2018.1432030. Epub 2018 Jan 30. PMID 29381390
- [Background] Tong, A. Y., & Man, D. W. (2002). The validation of the Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living Scale for institutionalized elderly persons. OTJR: Occupation, Participation and Health, 22(4), 132-142.
- [Background] Trambaiolli LR, Cassani R, Mehler DMA, Falk TH. Neurofeedback and the Aging Brain: A Systematic Review of Training Protocols for Dementia and Mild Cognitive Impairment. Front Aging Neurosci. 2021 Jun 9;13:682683. doi: 10.3389/fnagi.2021.682683. eCollection 2021. PMID 34177558
- [Background] Trambaiolli LR, Kohl SH, Linden DEJ, Mehler DMA. Neurofeedback training in major depressive disorder: A systematic review of clinical efficacy, study quality and reporting practices. Neurosci Biobehav Rev. 2021 Jun;125:33-56. doi: 10.1016/j.neubiorev.2021.02.015. Epub 2021 Feb 12. PMID 33587957
- [Background] van der Kolk BA, Hodgdon H, Gapen M, Musicaro R, Suvak MK, Hamlin E, Spinazzola J. A Randomized Controlled Study of Neurofeedback for Chronic PTSD. PLoS One. 2016 Dec 16;11(12):e0166752. doi: 10.1371/journal.pone.0166752. eCollection 2016. PMID 27992435
- [Background] Wager TD, Davidson ML, Hughes BL, Lindquist MA, Ochsner KN. Prefrontal-subcortical pathways mediating successful emotion regulation. Neuron. 2008 Sep 25;59(6):1037-50. doi: 10.1016/j.neuron.2008.09.006. PMID 18817740
- [Background] Wang SY, Lin IM, Fan SY, Tsai YC, Yen CF, Yeh YC, Huang MF, Lee Y, Chiu NM, Hung CF, Wang PW, Liu TL, Lin HC. The effects of alpha asymmetry and high-beta down-training neurofeedback for patients with the major depressive disorder and anxiety symptoms. J Affect Disord. 2019 Oct 1;257:287-296. doi: 10.1016/j.jad.2019.07.026. Epub 2019 Jul 5. PMID 31302517
- [Background] Wu, C. H., & Yao, G. (2006). Analysis of factorial invariance across gender in the Taiwan version of the Satisfaction with Life Scale. Personality and Individual Differences, 40(6), 1259-1268.
- [Background] Yeung MK, Lee TL, Chan AS. Frontal lobe dysfunction underlies the differential word retrieval impairment in adolescents with high-functioning autism. Autism Res. 2019 Apr;12(4):600-613. doi: 10.1002/aur.2082. Epub 2019 Feb 13. PMID 30758144
- [Background] Yeung MK, Lee TL, Chan AS. Right-lateralized frontal activation underlies successful updating of verbal working memory in adolescents with high-functioning autism spectrum disorder. Biol Psychol. 2019 Nov;148:107743. doi: 10.1016/j.biopsycho.2019.107743. Epub 2019 Aug 22. PMID 31445997
- [Background] Yeung MK, Lee TL, Chan AS. Depressive and anxiety symptoms are related to decreased lateral prefrontal cortex functioning during cognitive control in older people. Biol Psychol. 2021 Nov;166:108224. doi: 10.1016/j.biopsycho.2021.108224. Epub 2021 Nov 14. PMID 34785277
- [Background] Yeung MK, Lee TL, Chan AS. Negative mood is associated with decreased prefrontal cortex functioning during working memory in young adults. Psychophysiology. 2021 Jun;58(6):e13802. doi: 10.1111/psyp.13802. Epub 2021 Mar 4. PMID 33665829
- [Background] Yeung MK, Sze SL, Woo J, Kwok T, Shum DH, Yu R, Chan AS. Altered Frontal Lateralization Underlies the Category Fluency Deficits in Older Adults with Mild Cognitive Impairment: A Near-Infrared Spectroscopy Study. Front Aging Neurosci. 2016 Mar 29;8:59. doi: 10.3389/fnagi.2016.00059. eCollection 2016. PMID 27065857
- [Background] Yeung MK, Sze SL, Woo J, Kwok T, Shum DH, Yu R, Chan AS. Reduced Frontal Activations at High Working Memory Load in Mild Cognitive Impairment: Near-Infrared Spectroscopy. Dement Geriatr Cogn Disord. 2016;42(5-6):278-296. doi: 10.1159/000450993. Epub 2016 Oct 27. PMID 27784013
- [Background] Yochim, B. P., Mueller, A. E., June, A., & Segal, D. L. (2010). Psychometric properties of the geriatric anxiety scale: comparison to the beck anxiety inventory and geriatric anxiety inventory. Clinical Gerontologist, 34(1), 21-33.
- [Background] Zilverstand A, Sorger B, Sarkheil P, Goebel R. fMRI neurofeedback facilitates anxiety regulation in females with spider phobia. Front Behav Neurosci. 2015 Jun 8;9:148. doi: 10.3389/fnbeh.2015.00148. eCollection 2015. PMID 26106309

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT05936697/Prot_SAP_000.pdf